CLINICAL TRIAL: NCT05285449
Title: Influence of Cannabidiol on Glucose Tolerance and The Gut Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Bell (Other)
Collaborators: Caliper Foods (Unknown)
Responsible Party: Sponsor-Investigator, Christopher Bell, Associate Professor, Colorado State University
Organization: Colorado State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2065
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: Double-Blind random assignment to either placebo or active CBD (2 x 30 mg daily)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The CBD and placebo formulations are prepared, bottled, and coded by Caliper Foods. The participants will receive a coded bottle to consume of the different formulations of CBD and placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Supplement: Cannabidiol (CBD) powder formulation (Active Comparator): T-P-S-10 Caliper powder - 30 mg CBD in the form of 300 mg of 10% CBD isolate
  Interventions: Dietary Supplement: Cannabidiol (CBD) powder formulation
- Dietary Supplement: CBD matching Placebo (Placebo Comparator): Matching Placebo
  Interventions: Dietary Supplement: Matching Placebo Cannabidiol (CBD) powder formulation

INTERVENTIONS:
Dietary Supplement: Cannabidiol (CBD) powder formulation — 30 mg CBD in the form of 300 mg of 10% CBD isolate
  Other Names: T-P-S-10 Caliper powder
  Arms: Dietary Supplement: Cannabidiol (CBD) powder formulation
Dietary Supplement: Matching Placebo Cannabidiol (CBD) powder formulation — Matching Placebo
  Arms: Dietary Supplement: CBD matching Placebo

SUMMARY:
While many empirical projects have described multiple potential health benefits of CBD, the potential for CBD to provide protection against the development of diabetes via favorable modification of the gut microbiota has received relatively less attention. We hope to learn if CBD can improve glucose tolerance and the gut microbiota, and if these two improvements might be related.

DETAILED DESCRIPTION:
More than 122 million Americans have diabetes, or its precursor, pre-diabetes. The clinical and public health implications are not trivial as diabetes is the leading cause of blindness and non-traumatic amputation; it is closely associated with vascular disease and premature death, and people with diabetes are at greater risk of serious and fatal complications associated with Covid-19. The defining feature of diabetes is dysfunctional regulation of blood glucose (blood sugar). Although numerous factors contribute to the development of type 2 diabetes, the gut microbiota has recently emerged as an important regulator of glucose homeostasis. Imbalances in the microbiota can lead to intestinal inflammation and loss of gut barrier integrity, which in turn activates inflammatory cascades outside of the gut that can precipitate development of metabolic dysfunction. Changes in the gut microbiota can also alter proportions of microbial metabolites such as secondary bile acids and short chain fatty acids, which have been shown to influence host metabolism. Diet is one of the most important modifiers of the gut microbiota and several plant-based chemicals have been shown to exert beneficial effects on its composition and function. Cannabis sativa L., which produces a suite of phytochemicals, referred to collectively as cannabinoids, has also been shown in epidemiologic studies to exert beneficial effects on glucose regulation. These effects may be, in part, due to interactions with the gut microbiota. The focus of this project is cannabidiol (often abbreviated as CBD). CBD is not marijuana. CBD is not cannabis. CBD is a bioactive phytochemical that is present in the plant Cannabis sativa; it has no psychoactive properties. Over recent years CBD has garnered considerable attention on account of its potential medicinal properties. There is increasing evidence that CBD may have therapeutic and/or preventative effects pertinent to cancer, cardiovascular disease, anxiety, and most relevant to the current proposal, diabetes and the gut microbiota. The aim of the proposed study is to evaluate the influence of short-term CBD on glucose tolerance and the gut microbiota. Hypothesis: compared with daily ingestion of a placebo, 4-weeks daily ingestion of CBD will improve glucose tolerance and favorably modify the gut microbiota towards a more anti-inflammatory profile.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Weight more than 110 pounds
* Have a Body Mass Index greater than or equal to 25 kilograms/squared meters
* Free of gastrointestinal or metabolic diseases
* Sedentary (less than 150 minutes of moderate-intensity exercise per week during the previous 3 months)

Exclusion Criteria:

* Less than 18 years of age
* Pregnant or breastfeeding
* Have known food allergies
* Have been diagnosed with any autoimmune disorders or with compromised immune function
* Celiac disease
* Inflammatory bowel diseases
* Gastrointestinal cancers
* Diabetes
* Human Immunodeficiency Virus
* Adverse reaction to ingesting CBD oils, or CBD containing food products
* Taking any of the following medications will be excluded as these may have negative interactions with CBD:
* steroids,
* 3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitors,
* calcium channel blockers,
* antihistamines,
* human immunodeficiency virus antivirals
* immune modulators,
* benzodiazepines,
* antiarrythmics,
* antibiotics,
* anesthetics,
* antipsychotics,
* antidepressants,
* anti-epileptics,
* beta blockers,
* coumadin (warfarin),
* proton pump inhibitors,
* non-steroidal anti-inflammatory drugs,
* angiotension II blockers,
* oral hypoglycemic agents,
* sulfonylureas.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Circulating blood glucose | Compared to baseline after 4 weeks of the intervention
  Measurements of circulating blood glucose during an Oral Glucose Tolerance Tests via a blood analyzer
Circulating blood insulin | Compared to baseline after 4 weeks of the intervention
  Measurements of circulating insulin during an Oral Glucose Tolerance Tests via a blood analyzer
Hepatic Insulin Extraction | Compared to baseline after 4 weeks of the intervention
  Measurements of C-Peptide concentration via ELISA Assays
Tissue oxygenation | Compared to baseline after 4 weeks of the intervention
  Measurement of tissue oxygenation via Near-Infrared Spectroscopy (NIRS)
Reactive hyperemia | Compared to baseline after 4 weeks of the intervention
  Measurement of reactive hyperemia via doppler ultrasound
Shannon and Faith's microbiota diversity scores in feces | Compared to baseline after 4 weeks of the intervention
  Assessed via 16s ribosomal ribonucleic acid microbial profiling
B-diversity scores for all fecal samples to assess clustering | Compared to baseline after 4 weeks of the intervention
  Assessed via 16s ribosomal ribonucleic acid microbial profiling
Differentially abundant microbiota in feces of collected during treatment | Compared to baseline after 4 weeks of the intervention
  Assessed via 16s ribosomal ribonucleic acid microbial profiling
Abundant microbiota to markers in feces | Compared to baseline after 4 weeks of the intervention
  Assessed via Linear discriminant analysis Effect Size algorithm
Human Granulocyte Macrophage Colony-Stimulating Factor | Compared to baseline after 4 weeks of the intervention
  Assessed via 13-plex human T-cell cytokine panel
Interferon gamma | Compared to baseline after 4 weeks of the intervention
  Assessed via 13-plex human T-cell cytokine panel
Interleukin 1 beta | Compared to baseline after 4 weeks of the intervention
  Assessed via 13-plex human T-cell cytokine panel
Interleukin 2 | Compared to baseline after 4 weeks of the intervention
  Assessed via 13-plex human T-cell cytokine panel
Interleukin 4 | Compared to baseline after 4 weeks of the intervention
  Assessed via 13-plex human T-cell cytokine panel
Interleukin 5 | Compared to baseline after 4 weeks of the intervention
  Assessed via 13-plex human T-cell cytokine panel
Interleukin 6 | Compared to baseline after 4 weeks of the intervention
  Assessed via 13-plex human T-cell cytokine panel
Interleukin 7 | Compared to baseline after 4 weeks of the intervention
  Assessed via 13-plex human T-cell cytokine panel
Interleukin 8 | Compared to baseline after 4 weeks of the intervention
  Assessed via 13-plex human T-cell cytokine panel
Interleukin 10 | Compared to baseline after 4 weeks of the intervention
  Assessed via 13-plex human T-cell cytokine panel
Interleukin 12 (p70) | Compared to baseline after 4 weeks of the intervention
  Assessed via 13-plex human T-cell cytokine panel
Interleukin 13 | Compared to baseline after 4 weeks of the intervention
  Assessed via 13-plex human T-cell cytokine panel
Tumor Necrosis Factor alpha | Compared to baseline after 4 weeks of the intervention
  Assessed via 13-plex human T-cell cytokine panel
High-sensitivity C-reactive protein | Compared to baseline after 4 weeks of the intervention
  Assessed via 13-plex human T-cell cytokine panel

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado State University, Dept. of Health and Exercise Science, Fort Collins, Colorado, United States